CLINICAL TRIAL: NCT03972553
Title: Parastomal Hernia Repair Utilizing the Retromuscular Sugarbaker Versus Keyhole Mesh Techniques: A Registry-Based Randomized Controlled Trial
Brief Title: Parastomal Hernia Repair Utilizing the Retromuscular Sugarbaker Versus Keyhole Mesh Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clayton Petro (Other)
Responsible Party: Sponsor-Investigator, Clayton Petro, Associate Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-398
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Parastomal Hernia
Keywords: Sugarbaker; keyhole; Open parastomal hernia repair

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugarbaker (Other): For the Sugarbaker group, the bowel will be brought through the peritoneum lateral to the edge of the retromuscular mesh and then draped over the mesh before bringing it through the anterior fascia medially.
  Interventions: Procedure: Sugarbaker technique for repairing parastomal hernia
- Keyhole (Other): For the Keyhole group the stoma will be taken down and rematured through a cruciate incision (keyhole)
  Interventions: Procedure: Keyhole technique for repairing parastomal hernia

INTERVENTIONS:
Procedure: Sugarbaker technique for repairing parastomal hernia — The bowel will be brought through the peritoneum lateral to the edge of the retromuscular mesh and then draped over the mesh before bringing it through the anterior fascia medially.
  Arms: Sugarbaker
Procedure: Keyhole technique for repairing parastomal hernia — The bowel will be brought through defects in the posterior rectus sheath or contiguous peritoneum, mesh, and anterior fascia.
  Arms: Keyhole

SUMMARY:
This will be a randomized controlled trial comparing the incidence of radiographic hernia recurrence 2 years after parastomal hernia repair utilizing the retro-muscular Sugarbaker technique compared to the retro-muscular keyhole mesh technique. The primary endpoint will be recurrence at two years. Secondary endpoints will be the incidence of mesh-related complications, all 30-day complication rates, and hospital length of stay. Patients eligible for the study will be 18 years or older with a parastomal hernia that requires open repair retromuscular repair without ostomy reversal as determined by one of five hernia surgeons who will participate in this study at the investigators' institution. All patients will be marked for a new stoma site preoperatively. Patients who have insufficient bowel length suitable for either technique will be excluded intraoperatively. Patients enrolled in the study will be entered in the Americas Hernia Society Quality Collaborative database by the attending surgeon. The database houses patient demographics, medical comorbidities, operative details, and postoperative outcomes - all entered by the attending surgeon.

DETAILED DESCRIPTION:
Recent estimates approximate that 120,000 ostomies are created yearly, with an overall prevalence greater than 800,000. Parastomal hernia formation is the most common complication thereof, as most reviews acknowledge a rate of 50%, which increases to 75% for patients with a waist circumference >100cm. As patients live longer and rates of obesity climb, the sequelae of parastomal hernias do as well, including difficulty fitting stoma appliances, parastomal skin breakdown, pain, and obstructive episodes - all negatively impacting the patient's quality of life and compelling them to seek repair.

Recent data from the Americas Hernia Society Quality Collaborative (AHSQC) - a quality improvement hernia registry of surgeon-entered patient demographics, operative details, and outcomes - found that only 22% of stomas were reversible at the time of their parastomal hernia operation.[7] So in the vast majority of cases, the surgeon must decide the optimal technique for repair in the presence of a persistent stoma. Decision-making includes open versus laparoscopic approaches, stoma re-siting versus leaving it in situ, use of mesh, and mesh orientation relative to the bowel. The same AHSQC analysis found that mesh is used in 94% of repairs, and almost 80% are repaired open, likely due to the need for repair of a concomitant midline incisional hernia that frequently exists. As a high-volume hernia center, the investigators' preference has been to perform an open retromuscular repair with a transversus abdominis release (TAR) and retromuscular mesh placement, allowing for reinforcement of the midline, stoma, and prior stoma site if the stoma was re-sited. The stoma can be brought through a keyhole incision in the retromuscular mesh. The investigators' hernia recurrence rate at just 13-months mean follow-up was previously found to be 11%. A more recent audit of parastomal hernia repairs among the investigators using the aforementioned "keyhole" technique with a minimum of 1-year follow-up found a 17% rate of radiographic recurrence and 33% "composite" recurrence rate - patients who feel a bulge, regardless of their radiographic results. Recently, Pauli et al. reported the results of a novel technique for parastomal hernia repair at the 2018 International Hernia Congress with exciting early results. The technique is similar to the investigators' approach with a bilateral transversus abdominis release and placement of a retromuscular mesh reinforcement. However, rather than bringing the stoma through a keyhole defect in the mesh, it is draped over the mesh in the retromuscular space akin to a Sugarbaker repair offsetting the defect in the mesh and the fascia. Six surgeons reported their results of 44 patients with a mean follow-up of 10 months, with a 4.5% (n=2) recurrence rate, with no reports of mesh erosion or stoma necrosis. Given the excellent early results of this novel approach, the investigators hypothesize that the retromuscular Sugarbaker technique would dramatically reduce hernia recurrence compared to the traditional keyhole repair.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to give informed consent
* Patient has one parastomal hernia
* Patient is willing to undergo mesh-based repair
* Patient is considered eligible to undergo open retromuscular repair without ostomy reversal
* The patient can tolerate general anesthesia
* Repair being performed in an elective situation

Exclusion Criteria:

* The subject is <18 years of age
* Patient has more than one stoma
* The patient is unable to give informed consent
* Patient is not willing to undergo mesh-based repair due to any reason
* Patient not eligible for open retromuscular repair without ostomy reversal
* Patient is unable to tolerate general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Radiographic hernia recurrence 2 years after parastomal hernia repair | Two years after the last surgery
  To compare the incidence of radiographic hernia recurrence 2 years after parastomal hernia repair utilizing a retromuscular Sugarbaker technique compared to the retromuscular keyhole mesh technique.

SECONDARY OUTCOMES:
Incidence of mesh-related complications | Two years after the last surgery
  To compare the incidence of mesh-related complications between the two study groups.
30-day complication rates | 30 days after the last surgery
  To compare all 30-day complication rates for the two study groups.
Hospital length-of-stay | An average of 1 week after the last surgery
  To compare hospital length-of-stay for the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Petro, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Abdominal Core Health, Cleveland, Ohio, United States

REFERENCES:
- [Background] Turnbull GB. Ostomy statistics: the $64,000 question. Ostomy Wound Manage. 2003 Jun;49(6):22-3. No abstract available. PMID 12874481
- [Background] Hotouras A, Murphy J, Thaha M, Chan CL. The persistent challenge of parastomal herniation: a review of the literature and future developments. Colorectal Dis. 2013 May;15(5):e202-14. doi: 10.1111/codi.12156. PMID 23374759
- [Background] Carne PW, Robertson GM, Frizelle FA. Parastomal hernia. Br J Surg. 2003 Jul;90(7):784-93. doi: 10.1002/bjs.4220. PMID 12854101
- [Background] De Raet J, Delvaux G, Haentjens P, Van Nieuwenhove Y. Waist circumference is an independent risk factor for the development of parastomal hernia after permanent colostomy. Dis Colon Rectum. 2008 Dec;51(12):1806-9. doi: 10.1007/s10350-008-9366-5. Epub 2008 May 16. PMID 18483825
- [Background] Gavigan T, Stewart T, Matthews B, Reinke C. Patients Undergoing Parastomal Hernia Repair Using the Americas Hernia Society Quality Collaborative: A Prospective Cohort Study. J Am Coll Surg. 2018 Oct;227(4):393-403.e1. doi: 10.1016/j.jamcollsurg.2018.07.658. Epub 2018 Aug 4. PMID 30081081
- [Background] Timmermans L, Deerenberg EB, Lamme B, Jeekel J, Lange JF. Parastomal hernia is an independent risk factor for incisional hernia in patients with end colostomy. Surgery. 2014 Jan;155(1):178-83. doi: 10.1016/j.surg.2013.06.014. Epub 2013 Nov 12. PMID 24238119
- [Background] Raigani S, Criss CN, Petro CC, Prabhu AS, Novitsky YW, Rosen MJ. Single-center experience with parastomal hernia repair using retromuscular mesh placement. J Gastrointest Surg. 2014 Sep;18(9):1673-7. doi: 10.1007/s11605-014-2575-4. Epub 2014 Jun 19. PMID 24944155
- [Derived] Maskal SM, Ellis RC, Fafaj A, Costanzo A, Thomas JD, Prabhu AS, Krpata DM, Beffa LRA, Tu C, Zheng X, Miller BT, Rosen MJ, Petro CC. Open Retromuscular Sugarbaker vs Keyhole Mesh Placement for Parastomal Hernia Repair: A Randomized Clinical Trial. JAMA Surg. 2024 Sep 1;159(9):982-989. doi: 10.1001/jamasurg.2024.1686. PMID 38865142
- [Derived] Miller BT, Krpata DM, Petro CC, Beffa LRA, Carbonell AM, Warren JA, Poulose BK, Tu C, Prabhu AS, Rosen MJ. Biologic vs Synthetic Mesh for Parastomal Hernia Repair: Post Hoc Analysis of a Multicenter Randomized Controlled Trial. J Am Coll Surg. 2022 Sep 1;235(3):401-409. doi: 10.1097/XCS.0000000000000275. Epub 2022 Aug 10. PMID 35588504
- [Derived] Miller BT, Thomas JD, Tu C, Costanzo A, Beffa LRA, Krpata DM, Prabhu AS, Rosen MJ, Petro CC. Comparing Sugarbaker versus keyhole mesh technique for open retromuscular parastomal hernia repair: study protocol for a registry-based randomized controlled trial. Trials. 2022 Apr 4;23(1):251. doi: 10.1186/s13063-022-06207-x. PMID 35379311